CLINICAL TRIAL: NCT07309510
Title: Effectiveness of a Counseling Program on Exclusive Breastfeeding Rates in a Primary Care Center in A Coruña.Randomized Controlled Clinical Trial
Brief Title: Effectiveness of a Counseling Program on Exclusive Breastfeeding Rates in a Primary Care Center
Acronym: ALM-AP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Profesor Novoa Santos (Other)
Responsible Party: Principal Investigator, Yolanda Sánchez Suárez, Nurse specialist in Pediatric Nursing, Fundacion Profesor Novoa Santos
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025/235; 2025/235 (Other: Comité de Ética de la Investigación de A Coruña- Ferrol)
Record Dates: First submitted 2025-11-19; First posted 2025-12-30 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Growth & Development; Breastfeeding Satisfaction; Breastfeeding Consultancy Training; Breastfeeding Duration; Breastfeeding After Discharge From Hospital Following Childbirth, Yes/no; Breastfeeding, Exclusive; Breastfeeding Attitude; Breastfeeding Support System; Breastfeeding Rate; Breastfeeding Outcomes
Keywords: Breastfeeding; Infant; Human Milk; Health Education; Primary Health Care; Postpartum Period
MeSH Terms: conditions — Breast Feeding; Health Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional care (No Intervention): Conventional care within the Child Health Program (SERGAS) The health program includes 5 appointments with the Pediatric Specialist doctor and the Pediatric Specialist nurse in the first 6 months of life. These appointments will take place at 7-15 days, at 1 month, at 2 months, at 4 months, and at 6 months of age.
- breastfeeding counseling (Experimental)
  Interventions: Behavioral: breastfeeding counseling

INTERVENTIONS:
Behavioral: breastfeeding counseling — The intervention group will receive, in addition to the indicated conventional care, 4 scheduled breastfeeding counseling appointments, the first of which will take place within the first 72 hours after hospital discharge following birth. As part of the breastfeeding counseling, the Latch scale will be used to observe and assess breastfeeding sessions, the breastfeeding self-efficacy scale-short (BSES-SF) to evaluate breastfeeding self-efficacy, the Visual Analogue Scale (VAS) to evaluate pain related to breastfeeding, and the breastfeeding clinical record form from the World Health Organization (WHO). Training will be provided to the mother and family on pre-selected breastfeeding topics. Mothers will be able to contact the IP nurse by phone daily on demand from 10 a.m. to 3 p.m.
  Arms: breastfeeding counseling

SUMMARY:
Introduction: Evidence supports that exclusive breastfeeding (EBF) is the most beneficial method of infant feeding up to 6 months of age. The practice confers numerous advantages for the infant and the mother. Many breasfeeding are abandoned early due difficulties experienced after dischargue and after returning to work. Development specific early breastfeeding support programs in the community is necessary to avoid unwanted abandonment.

Objective: To analyse the differences in BF rates at six month of birth in healthy full-term newborns between the study groups.

Methodology: Pilot study of a randomised clinical trial carried out in a Paediatric Nursing clinic at the Ventorrillo Health Centre in A Coruña. The study population will be mothers of healthy full-term newborns who wish to give BF at the time of delivery and whose reference health centre is the one of the study. The mother- newborn dyads in the control group (CG) will receive the usual care described in the child health Program of the Galician Health Service, and the dyads included in the intervention group (IG) will also receive specific advice on breastfeeding during the first 6 months of life. A study sample of 80 participants is estimated for each group. The study will be approved by the Research Ethics Committee of A Coruña-Ferrol. The variables under study will be collected in a data collection notebook for later statistical analysis. A significant value of p < 0.05 being considered.

ELIGIBILITY:
Inclusion Criteria:

* Mothers who express a desire to breastfeed during a follow-up consultation with the Obstetric and Gynecological Nursing specialist at 36 weeks of gestation.
* Mothers who plan to give birth at HMI of CHUAC, referred from the C.S. Ventorrillo.
* Women who are fluent in Spanish or Galician.

Exclusion Criteria:

* Maternal age under 18 years - Maternal use of drugs or medication that prevent breastfeeding .
* Maternal infection with HIV or Human T-cell Leukemia Virus.
* Mothers of newborns with cow's milk protein allergy, galactosemia, or congenital primary lactase deficiency.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Rate of exclusive breastfeeding at 6 months of age of the newborn | From birth up to 6 months of the infant's life
  The practice of feeding the infant exclusively with breast milk from 0 to 5 months (without giving any other food or drink, not even water). Nursing by a wet nurse, feeding with expressed breast milk, and feeding with breast milk from donors are also considered breastfeeding.

SECONDARY OUTCOMES:
Number of participants with exclusive breastfeeding at 15 days, one month, and three months of the newborn's life. | At 15 days, one month, and three months of the newborn's life.
  Defined as the practice of feeding the infant exclusively with breast milk (without giving any other food or drink, not even water). Breastfeeding by a wet nurse, feeding with expressed breast milk, and feeding with donor breast milk are also considered breastfeeding.
Number of participants with recovery to birth weight | At 15 days and one month of age
  The infant regains the weight with which they were born
Grams of daily weight gain | At 15 days, 1 month, 2 months, 4 months and 6 months of the infant's life
  Grams of weight gained per day since the previous weight check.
Age of introduction of complementary feeding | From birth to 6 months of age
  Age of the infant at which complementary feeding is started in both study groups.
Number of Hospital admissions by the newborn | From birth to 6 months of age
  Hospital admissions by the newborn in both study groups.
Number of emergency department visits by the newborn | From birth to 6 months of age
  number and reason for emergency department visits by the newborn in both study groups.
Number of visits by the pediatric nurse specialist | Until completion of the study (6 months after birth)
  Number and reason for visits by the pediatric nurse specialist in both study groups.
Number of visits to the specialist nurse in Obstetric-Gynecological Nursing | Until completion of the study (6 months after birth)
  Number of visits to the specialist nurse in Obstetric-Gynecological Nursing
Days after birth of cessation of breastfeeding | Until completion of the study (6 months after birth)
  Days of the infant's life when the last breastfeeding is administered
Reasons reasons given by the mother in an interview for breastfeeding abandonment | 6 months after birth or when the mother abandons the study
  Reasons for breastfeeding discontinuation among the study groups.
Score on the validated scale of impact of support networks in breastfeeding | 6 months after birth or when the mother abandons the study
  Score on the validated scale of impact of support networks in breastfeeding Validated scale of the impact of support networks on breastfeeding. Composed of 12 items, self-administered. Mothers must indicate their level of agreement or disagreement with the statements using a 5-point Likert scale. The maximum score is 60 points and the minimum is 12 points. A higher score indicates a greater degree of satisfaction or perceived quality among users of breastfeeding support services.
Score of Maternal Breastfeeding Evaluation Scale (MBFES-E) | 6 months after birth or when the mother abandons the study
  Score on the Spanish version of the Maternal Breastfeeding Evaluation Scale (MBFES-E). A 5-point Likert-type scale is used in which the participant rates their level of agreement with the item statement (1: strongly disagree to 5: strongly agree). The final score on the scale will range from 30 to 150 and is interpreted such that a higher score indicates greater satisfaction with the breastfeeding experience.

CONTACTS AND LOCATIONS:
Overall Officials: Yolanda Sánchez Suárez, Principal Investigator — Servicio Gallego de Salud; Carmen Neri Fernández Pombo, PhD, Principal Investigator — Servicio Gallego de Salud. Instituto de Investigación Biomédica de A Coruña.; Javier Muñíz García, PhD, Study Director — Universidade de A Coruña
Locations (1):
- Centro de Salud de O Ventorrillo, A Coruña, Galicia, Spain

IPD SHARING:
Plan to Share IPD: No